CLINICAL TRIAL: NCT04810065
Title: SingStrong: Strong Lungs Through Song
Brief Title: SingStrong: Strong Lungs Through Song - Long COVID-19 Study
Acronym: ss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Roisin Cahalan, Senior Lecturer Physiotherapy, University of Limerick
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SingStrong
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Long Covid
Keywords: Singing; Disordered breathing; Covid-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SingStrong for Pulmonary Fibrosis (Other): This arm of the project explores Singing as an intervention for people suffering from Pulmonary Fibrosis specifically.
  It is a 10 week programme. All other aspects of the intervention are the same in terms of delivery and length of classes.
  Different outcome measures, namely the St Georges Respiratory Questionnaire is used in this trial. This is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
  Interventions: Other: SingStrong: Strong lungs through Song

INTERVENTIONS:
Other: SingStrong: Strong lungs through Song — Participants who have been clinically diagnosed with Covid-19 and who continue to suffer residual adverse effects on the lung health will be invited to participate in the study.
  The intervention will involve biweekly hour-long breathing and singing classes that are designed to correct dis-ordered breathing, and retrain the principal muscles of respiration.
  Pre and post evaluation of participant bio-psychosocial health and wellness will be conducted. Triangulation of data using focus groups and individual interviews will be conducted after conclusion of the intervention,

SUMMARY:
Evidence is emerging that many individuals who recover from Covid-19 are experiencing a range of residual problems. These include fatigue, pain, reduced exercise tolerance and breathing issues. This study includes participants who are experiencing problems with their lungs such as breathing difficulties, shortness of breath, and/or reduced exercise tolerance. The intervention is a twice weekly singing and breathing retraining intervention conducted over ten weeks. A range of self-report questionnaire measures will evaluate the efficacy of the intervention in addressing these problems. Focus groups and individual interviews will also be used to gather information on the impact and acceptability of the programme.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Previous clinical diagnosis of Covid-19
* Ongoing issues with any or all of: Shortness of breath, disordered breathing, reduced exercise tolerance
* Good written and spoken English language

Exclusion Criteria:

* Lack of a confirmed Covid-19 diagnosis
* Currently undergoing a similar singing or breathing retraining intervention
* No residual problems from a confirmed case of Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Covid-19 Yorkshire Rehab Screen (C19YRS) | 12 weeks
  The C19YRS was developed as a screening tool to monitor long-term symptoms due to Covid-19. The screening tool covers 19 items which combines yes/no answers and an 11 point ordinal scale (0-10) where a higher score denotes increased symptom severity.

SECONDARY OUTCOMES:
DePaul Symptom Questionnaire - Short Form DSQ - SF | 12 weeks
  The DPSQ -SF assesses key symptoms of ME/Chronic Fatigue Syndrome such as fatigue, post-exertional malaise, sleep, pain, neurological/cognitive impairments and autonomic, neuroendocrine and immune symptoms. At each item, participants have to rate the frequency and severity of the symptom on a scale from 0 to 4. A higher score denotes increased symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Roisin Cahalan, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No